CLINICAL TRIAL: NCT07361406
Title: SweetSpot - The Effect of Non-nutritive Sweeteners on Glucose Regulation, Gut Microbiome, and Gut Hormone Secretion in Healthy Adults: a Fully Controlled Cross-over Intervention Study
Brief Title: SweetSpot - The Effect of Non-nutritive Sweeteners on Health
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Food & Biobased Research - Wageningen UR (Unknown); TKI Agri & Food (Unknown); The Magnum Ice Cream Company (Unknown); Tate & Lyle (Industry); Symrise AG (Unknown); American Beverage Association (Other); Yildiz Holding (Unknown)
Responsible Party: Principal Investigator, Monica Mars, Dr. Ir. Monica Mars, Wageningen University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: NL010297
Record Dates: First submitted 2026-01-13; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Healthy Adult
Keywords: glucose metabolism; gut microbiome; gut hormones; non-nutritive sweeteners
MeSH Terms: interventions — Diet; Non-Nutritive Sweeteners

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NNS / no-NNS (Other): In this arm, participants will first receive the NNS diet, and the no-NNS diet in the second study period.
  Interventions: Other: Diet with non-nutritive sweeteners; Other: Diet without non-nutritive sweeteners
- No-NNS / NNS (Other): In this arm, participants will first receive the no-NNS diet, and the NNS diet in the second study period.
  Interventions: Other: Diet with non-nutritive sweeteners; Other: Diet without non-nutritive sweeteners

INTERVENTIONS:
Other: Diet with non-nutritive sweeteners — Fully controlled diet with added mixture of non-nutritive sweeteners. The mixture consist of 6 different non-nutritive sweeteners: acesulfame-K, aspartame, cyclamate, saccharin, sucralose, and rebaudioside A (stevia).
Other: Diet without non-nutritive sweeteners — Fully controlled diet without any non-nutritive sweeteners added.

SUMMARY:
The aim of the study is to investigate the effect of non-nutritive sweeteners on glucose regulation. Secondary objectives are to investigate the effect of NNS on gut microbiome, gut hormone secretion, sweet taste sensitivity and preference, and the excretion of NNS in urine.

DETAILED DESCRIPTION:
Sugar intake has increased over the years, simultaneously with the prevalence of overweight and obesity. To decrease sugar intake, consumption of non-nutritive sweeteners (NNS) has increased and opinions on its use remain divided. A fully controlled dietary intervention using a NNS mixture and dose that is similar to real-life intake, is therefore necessary to advance our understanding of the potential effects of NNS on glucose regulation, gut microbiome, and gut hormone secretion under real-life conditions.

The aim of this study is to investigate the effect of non-nutritive sweeteners on glucose regulation. Secondary objectives are to investigate the effect of NNS on gut microbiome, gut hormone secretion, sweet taste sensitivity and preference, and the excretion of NNS in urine.

To do this, a single blind, fully controlled dietary intervention with a cross-over design will be performed. The study will consist of 2x8 weeks of intervention, with a washout of > 6 weeks in between. The study population will be 60 healthy adults aged 45-79, with a BMI between 20-35 kg/m2.

The study will consist of a fully controlled diet of two 8-week intervention periods (2 weeks run-in + 6 weeks intervention). The diets differ in the presence of non-nutritive sweeteners (NNS): NNS-diet versus non-NNS diet, where additional NNS are added to the NNS-diet.

The primary outcome measure will be the within person difference in blood glucose incremental area under the curve following a 75 g glucose tolerance test between the NNS diet and the non-NNS diet. Secondary outcome measures are the effect of NNS on Matsuda index, insulin response, blood lipid profile, and gut hormone secretion will be determined. The effect of NNS on small- and large intestinal microbiome will be investigated by a change in composition, functionality, and short chain fatty acid content. The effect of NNS on sweet taste sensitivity, preference, and liking will be investigated, as well as the excretion of NNS in urine and saliva.

The total time invested by participants is around 85 hours. Participants are restricted for 16 weeks in their eating habits, since they follow a fully controlled diet prepared by the research facility. Participants will visit the research facility in total 38 times. In total, ~ 603 mL of blood will be drawn by experienced nurses over the entire RCT (>6 month period). During DEXA scans, participants will receive a total of about 0.006 mSv of radiation.

Invasive measurements that participants can experience as burden are collection of faecal and urine samples, and finding back the Simba capsules in the stool. Non-invasive measurements for participants are wearing the CGM, wearing the ActiGraph, consuming the blue cakes, and performing sensory tests.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-79 years;
* BMI of 20-35 kg/m2;
* Having veins suitable for placement of a venflon catheter.

Exclusion Criteria:

* Diseases or prior surgeries affecting the stomach, liver, kidneys or intestines (allowed i.e. appendectomy);
* Cardiovascular diseases (e.g. heart failure) or cancer (e.g. non-invasive skin cancer allowed);
* Diagnosed with type 1 or type 2 diabetes;
* Drug treated thyroid diseases (well substituted hypothyroidism is allowed for inclusion);
* HbA1c level >6.5% (>48 mmol/mol), as measured during the screening visit;
* Anaemia defined as Hb concentrations <8.5 mmol/L for men and <7.5 mmol/L for women via finger prick;
* Regular use of/receiving medication interfering with research outcomes (as judged by research physician), such as use of glucose lowering drugs, insulin, or use of medication that impacts the gastro-intestinal system;
* Use of antibiotics over the last 3 months before study start;
* Donated blood within 2 months prior to the screening;
* Food allergies, intolerances (including lactose/gluten intolerance) for products used in the study design and/or dietary restrictions interfering with the study (including special diets and eating disorders);
* Followed a diet that can interfere with the study outcomes within 1 month prior to the screening (e.g. ketogenic, sugar free, carbohydrate free);
* Not willing to eat all products in the study diet, including eggs and dairy. Vegetarian is possible;
* Not willing to consume non-nutritive sweeteners;
* Not willing to quit the use of supplements that can interfere with the study outcomes (e.g. pre- or probiotics).
* Intention to change the intensity of exercise during the study period or planning to join a intensive sport event (e.g. marathon or triathlon);
* Intention to lose or gain weight;
* Working night shifts regularly;
* Smoking regularly
* Use of soft and/or hard drugs (cannabis included);
* Abuse of alcohol (defined as >14 glasses (women) or >21 glasses (men) of alcoholic beverages per week);
* Being pregnant or lactating or planning to become pregnant;
* Inability to understand study information and/or communicate with staff;
* Participation in another study that involves an intervention within two months prior to the intervention;
* Working or doing a thesis/internship at the division of Human Nutrition & Health, or the Food, Health & Consumer Research group of Wageningen Food & Biobased Research.

Ages: 45 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-11-26 (Estimated); Study Completion 2026-11-26 (Estimated)

PRIMARY OUTCOMES:
Difference in change in 2h iAUC glucose after 6 weeks between the intervention and the control. | Week 2 and week 8 in both intervention periods (4 times in total)
  The primary outcome measure is the difference in change in iAUC of blood glucose levels following a 2-hour oral glucose tolerance test (OGTT) after six weeks between the intervention period and the control period.

SECONDARY OUTCOMES:
Matsuda index | Week 2 and week 8 in both intervention periods (4 times in total)
  Matsuda index after an OGTT
Fasting blood glucose | Baseline & 2 times per intervention period (week 2 and week 8). 5 times in total.
  Fasting blood glucose
Fasting blood insulin | Baseline & 2 times per intervention period (week 2 and week 8). 5 times in total.
  Fasting blood insulin
Postprandial insulin response | Week 2 and 8 in both intervention periods (4 times in total).
  2-hour iAUC blood insulin during OGTT
Postprandial glucose response after a breakfast | Week 7 in both study periods (2 times in total)
  Postprandial blood glucose responses (PPGR) following specific meals measured by CGM.
Blood lipid profile | Baseline & 2 times per intervention period (week 2 and week 8). 5 times in total.
  All circulating blood lipids, including all cholesterol types, triglycerides, and free fatty acids (FFAs).
Gut microbiota composition | Average of three samples per timepoint. Measured at baseline & 2 times per intervention period (week 2 and week 8). 15 samples over 5 timepoints in total.
  Microbiota composition in faeces
Gut microbiota function | Average of three samples per timepoint. Measured at baseline & 2 times per intervention period (week 2 and week 8). 15 samples over 5 timepoints in total.
  Microbiota functionality measured in faeces
Microbial metabolites | Average of three samples per timepoint. Measured at baseline & 2 times per intervention period (week 2 and week 8). 15 samples over 5 timepoints in total.
  Microbial metabolites measured in faeces
Small intestinal microbiota composition | Week 7 of both intervention periods (2 times in total).
  Microbiota composition of the small intestine measured with Simba Capsules
Gastro-intestinal transit time | Baseline & week 7 of both intervention periods (3 times in total).
  Gastro-intestinal transit time measured with blue muffins.
Oral microbiome composition & function | Baseline & 2 times per intervention period (week 2 and week 8). 5 times in total.
  Oral microbiome composition & function measured in saliva
Postprandial GLP-1 secretion | Week 2 and 8 of both intervention periods (4 times in total).
  3-hour AUC of GLP-1 during an OGTT.
Postprandial GIP secretion | Week 2 and 8 of both intervention periods (4 times in total).
  3-hour AUC of GIP during an OGTT.
Sweetness-liker phenotype | Baseline & 2 times per intervention period (week 2 and week 8). 5 times in total.
  Sweetness-liker phenotype, with the sweetness liker test.
Sweetness preference & liking | Baseline & 2 times per intervention period (week 2 and week 8). 5 times in total.
  Sweetness preference & liking
Sweet taste sensitivity | Baseline & 2 times per intervention period (week 2 and week 8). 5 times in total.
  Sweet taste sensitivity
Sweet taste detection threshold | Baseline & 2 times per intervention period (week 2 and week 8). 5 times in total.
  Sweet taste detection threshold
Excretion of NNS in urine | Baseline, week 2 and week 8 in intervention period 1, and every two weeks in intervention period 2 (7 times in total).
  Excretion of NNS in urine
Excretion of NNS in saliva | Baseline & 2 times per intervention period (week 2 and week 8). 5 times in total.
  Excretion of NNS in saliva

OTHER OUTCOMES:
Anthropometrics | Baseline
  Measured as weight, height, waist circumference, and hip circumference
Body composition | Baseline & week 8 of both intervention periods (3 times in total).
  Body composition as measured by DEXA (Dual Energy X-ray Absorptiometry).
Habitual food intake | Baseline
  Habitual dietary intake assessment with a food frequency questionnaire (FFQ).
Physical activity level | Baseline.
  Physical activity level by the Short Questionnaire to Assess Health-enhancing physical activity (SQUASH).
Habitual NNS consumption | Baseline
  Habitual NNS consumption by questionnaire
Gastro-intestinal symptoms | Every week.
  Gastro-intestinal symptoms by GSRS questionnaire.
Satiety | Every week.
  Satiety questionnaire, adapted from the Control of Eating Questionnaire.
Genetic variation | Baseline
  Single Nucleotide Polymorphisms (SNPs) in genes relevant collected using buffycoat.

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University & Research, Wageningen, Gelderland, Netherlands